CLINICAL TRIAL: NCT00551941
Title: A Prospective Randomised Controlled Trial on the Use of BMP-7 (OP-1®) and Demineralised Bone Matrix in Tibial Non-union
Brief Title: A Prospective Randomized Controlled Trial on the Use of Bone Morphogenetic 7 (BMP-7) (OP-1®) and Demineralized Bone Matrix in Tibial Non-union
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment problems
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007/341
Record Dates: First submitted 2007-10-30; First posted 2007-11-01 (Estimated); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Non-union Diaphysary Tibial Fractures
MeSH Terms: interventions — Bone Morphogenetic Protein 7; Dopamine beta-Hydroxylase

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): non-union of diaphysary tibial fractures will be treated with allograft together with DBM
  Interventions: Procedure: allograft together with DBM
- 1 (Experimental): non-union of diaphysary tibial fractures will be treated with BMP-7 in adjunct to fresh frozen allograft
  Interventions: Procedure: BMP-7 in adjunct to fresh frozen allograft

INTERVENTIONS:
Procedure: BMP-7 in adjunct to fresh frozen allograft — non-union of diaphysary tibial fractures treated with BMP-7 in adjunct to fresh frozen allograft
  Arms: 1
Procedure: allograft together with DBM — non-union of diaphysary tibial fractures treated with allograft together with DBM
  Arms: 2

SUMMARY:
The researchers propose a prospective, randomised partially-blinded study to investigate the clinical and radiological outcome, effect on quality of life and socio-economic impact of non-union of diaphysary tibial fractures treated with BMP-7 in adjunct to fresh frozen allograft, in comparison to treatment with allograft together with DBM (demineralised bone matrix).

ELIGIBILITY:
Inclusion Criteria:

* Diaphysary tibial non-unions will be included (9 months after first surgery)
* Major surgery includes exchange nailing, bone grafting, internal fixation, amputation and soft-tissue coverage procedures, such as delayed primary closure and free flaps
* Surgery is classified as minor for removal of external fixator pins for local infection and removal of a static locking screw from intramedullary nails, a procedure known as dynamization
* ASA 1 and ASA 2
* Gap length/bone contact detected (1-5 cm): largest cortical gap in any radiographic incidence
* Subject or legal guardian is willing and able to understand, sign and date the study specific Patient Informed Consent, which has been approved by the Institutional Review Board
* Agrees to participate in post-operative evaluations and required rehabilitation regimen

Exclusion Criteria:

* Patients with known hypersensitivity to the active substance or collagen
* Gap more than 5 cm
* Immature skeleton
* Known auto-immune disease, including rheumatoid arthritis, systemic lupus erythematosus, scleroderma, Sjögren's syndrome and dermatomyositis/polymyositis
* Active infection on unhealed site or active systemic infection
* Non-healing resulting from pathological fractures, tumours or metabolic bone diseases
* Presence of tumour in vicinity of non-union
* Patients receiving chemotherapy, radiotherapy or immunosuppressant treatment or excessive steroids
* Patients with severely compromised soft tissue coverage or vascularisation at the non-union site, sufficient to impair bone healing
* Patients with congenital non-union
* Pregnancy and lactation
* Non-union of multiple bones interfering with walking
* Patients with neuromuscular diseases or conditions interfering normal weight bearing
* Patients who, judged by the surgeon, are candidates for just internal fixation alone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-10 (Actual); Primary Completion 2012-07-09 (Actual); Study Completion 2012-07-09 (Actual)

PRIMARY OUTCOMES:
X-ray evaluation | After 9 months
Change in VAS and LEFS scores | After 9 months

SECONDARY OUTCOMES:
Time of incapacity to work | Until ability to work
Change in SF-36 | After 4 years
Total socio-economic cost estimation | After 4 years
Repeated surgery (minor and major) | After 4 years
(Surgical) complications | After 4 years
Ability to bear weight (% of body weight) | After 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Rene Verdonk, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - AZ Sint Jan-Brugge, Bruges
  - University Hospital Ghent, Ghent